CLINICAL TRIAL: NCT03776942
Title: Synovial Chondrosarcoma: a Single Institution Experience
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: SynoChondroS
Record Dates: First submitted 2018-12-10; First posted 2018-12-17 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2018-12

CONDITIONS: Synovial Chondrosarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — tumor samples will be analysed by Dr. Dei Tos
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
single institution cases series review of histological, radiological and clinical data

DETAILED DESCRIPTION:
single institution cases series review of histological, radiological and clinical data. Investigators will retrieve from the archives of the Rizzoli institute all the cases with a histological diagnosis of synovial chondrosarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients treated at Rizzoli Institute from 01 January 1982 to 31 December 2017
* Diagnosis of synovial chondrosarcoma
* Age ≥ 18 years
* Histological slides / formalin-fixed paraffin-embedded tissue tumor (FFPE) blocks from archive available to perform the histology analysis
* Written informed consent prior to any study-specific analysis and/or data collection

Exclusion Criteria:

* Patients with histological diagnosis different from synovial chondrosarcoma

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and Female ≥ 18 years with diagnosis of synovial chondrosarcoma with histological slides/formalin-fixed paraffin-embedded tissue tumor blocks from archive available to perform the histology analysis
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
selection and review of cases of Synovial Chondrosarcoma | baseline (Day0)
  IDH1 and IDH2 analysis will be performed in order to better understand tumor characteristics and to identify the best therapeutic approach.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCC Rizzoli Orthopedic Institute, Bologna, Italy

REFERENCES:
- [Result] Ng VY, Louie P, Punt S, Conrad EU. Malignant Transformation of Synovial Chondromatosis: A Systematic Review. Open Orthop J. 2017 May 31;11:517-524. doi: 10.2174/1874325001711010517. eCollection 2017. PMID 28694891
- [Result] Biazzo A, Confalonieri N. Synovial chondrosarcoma. Ann Transl Med. 2016 Aug;4(15):280. doi: 10.21037/atm.2016.06.23. PMID 27570774
- [Result] Zamora EE, Mansor A, Vanel D, Errani C, Mercuri M, Picci P, Alberghini M. Synovial chondrosarcoma: report of two cases and literature review. Eur J Radiol. 2009 Oct;72(1):38-43. doi: 10.1016/j.ejrad.2009.05.029. Epub 2009 Jun 11. PMID 19523777
- [Result] Campanacci DA, Matera D, Franchi A, Capanna R. Synovial chondrosarcoma of the hip: report of two cases and literature review. Chir Organi Mov. 2008 Dec;92(3):139-44. doi: 10.1007/s12306-008-0062-3. Epub 2008 Dec 4. PMID 19057985
- [Result] Bertoni F, Unni KK, Beabout JW, Sim FH. Chondrosarcomas of the synovium. Cancer. 1991 Jan 1;67(1):155-62. doi: 10.1002/1097-0142(19910101)67:13.0.co;2-w. PMID 1985712

DOCUMENTS (1):
  • Study Protocol (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT03776942/Prot_000.pdf